CLINICAL TRIAL: NCT01686256
Title: A Multi-center Clinical Study to Evaluate the Safety and Efficacy of FolateScan (Technetium Tc 99m EC20) in Women With Suspected Ovarian or Endometrial Cancer
Brief Title: Safety and Efficacy of FolateScan (Technetium Tc 99m EC20) in Women With Suspected Ovarian or Endometrial Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Endocyte (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EC20.2
Record Dates: First submitted 2012-09-09; First posted 2012-09-18 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2012-09

CONDITIONS: Ovarian Cancer; Endometrial Cancer
Keywords: Ovarian Cancer; Endometrial Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms

ARMS (1):
- Tc 99m EC20 (Experimental): A Phase 1, multi-center, open-label, single-treatment group, baseline-controlled (for safety) study designed to verify product safety, determine optimal imaging time, gather efficacy data for the radioactive drug product (Technetium Tc 99m EC20), and assay masses for presence of folate receptors, in women with suspected ovarian or endometrial cancer. Twelve subjects will be enrolled, with a minimum of five malignant cases, as determined by histopathological evaluation.
  Interventions: Drug: Tc 99m EC20

INTERVENTIONS:
Drug: Tc 99m EC20 — Each subject will receive 1 mg of folic acid injected 1-3 minutes prior to administration of Technetium Tc 99m EC20.

SUMMARY:
A Multi-Center Clinical Study to Evaluate the Safety and Efficacy of FolateScan (Technetium Tc 99m EC20) in Women with Suspected Ovarian or Endometrial Cancer.

Phase I - The proposed indication for FolateScan is disease or pathological assessment of ovarian or endometrial masses.

DETAILED DESCRIPTION:
The study is designed to verify product safety, determine optimal imaging time, gather efficacy data for the radioactive drug product (Technetium Tc 99m EC20), and assay masses for presence of folate receptors, in women with suspected ovarian or endometrial cancer. Twelve subjects will be enrolled, with a minimum of five malignant cases, as determined by histopathological evaluation.

Women with a suspected ovarian or endometrial mass who either 1) have fixed, paraffin embedded tissue sample(s) available for immunohistochemical staining obtained from a previous pathological evaluation or 2) are scheduled for a procedure to obtain tissue for pathological evaluation that can be fixed and paraffin embedded for immunohistochemical staining are eligible for this study. The ovarian mass may be either an initial finding, e.g., found at a routine pelvic examination or to investigate symptoms, or the ovarian or endometrial mass may be a finding suspicious of recurrent or residual tumor at follow-up examination after surgical resection of confirmed ovarian or endometrial cancer. Patients may not be pregnant or breastfeeding at enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet the following eligibility requirements to be enrolled in the study.

  1. Subjects must be female, 18 years of age or older.
  2. Subjects must have suspected ovarian cancer or metastatic or recurrent ovarian or endometrial cancer with a known pelvic mass as diagnosed by ultrasound, MRI, or CT.
  3. Subjects either are scheduled to undergo a procedure to obtain tissue for pathological evaluation that can be fixed and paraffin embedded for immunohistochemical staining or have sufficient amounts of fixed, paraffin embedded tissue sample(s) available for immunohistochemical staining obtained from a previous pathological evaluation.
  4. Subjects must provide written informed consent prior to enrollment.
  5. Subjects must have kidney function with a creatinine value <2.0 mg/dL (within the previous 30 days).

Exclusion Criteria:

* Subjects must be excluded if any of the following conditions are present:

  1. Subject is pregnant or breast-feeding.
  2. Subject is simultaneously participating in another investigative drug study.
  3. Subject has completed the follow-up phase of any previous study less than 30 days prior to enrollment in this study.
  4. Subject is unable to tolerate conditions for radionuclide imaging.
  5. Subject has been administered another radiopharmaceutical that would interfere with the assessment of Technetium Tc 99m EC20.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2001-08; Primary Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James W. Fletcher, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Medical Center, Indianapolis, Indiana, United States